CLINICAL TRIAL: NCT03192488
Title: Effect of an H1 Receptor Antagonist on Exercise Performance in Hypoxia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Robert Chapman, Associate Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1702396373
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Hypoxia, Altitude
MeSH Terms: conditions — Altitude Sickness | interventions — Cetirizine; Altitude

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cetirizine/Hypoxia (Experimental): Subjects orally ingested 10 mg of Cetirizine 60 min before exercising in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  Interventions: Drug: Cetirizine; Other: Hypoxia
- Placebo/Normoxia (Placebo Comparator): Subjects orally ingested a 10 mg gelatin Placebo 60 min before exercising in a normoxic (room-air) environment (20.9% oxygen).
  Interventions: Drug: Placebo oral capsule
- Placebo/Hypoxia (Placebo Comparator): Subjects orally ingested a 10 mg Placebo 60 min before exercising in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  Interventions: Drug: Placebo oral capsule; Other: Hypoxia

INTERVENTIONS:
Drug: Cetirizine — Cetirizine tablet 10 mg
  Other Names: Zyrtec
  Arms: Cetirizine/Hypoxia
Drug: Placebo oral capsule — Gelatin placebo
  Arms: Placebo/Hypoxia; Placebo/Normoxia
Other: Hypoxia — Exposure to a 14.3% oxygen environment simulating an altitude of 3,000m/9,000ft
  Other Names: altitude, low-oxygen environment
  Arms: Cetirizine/Hypoxia; Placebo/Hypoxia

SUMMARY:
This study seeks to determine whether a simple, single intervention of Cetirizine / Zyrtec® use can improve exercise performance of active individuals when acutely exposed to altitude. For this project, healthy subjects will perform steady state and progressive work rate exercise, endurance performance time trials, and repeated sprint performance time trials in the laboratory at a simulated altitude of 3000m (9900ft) after dosing with 10 mg of Cetirizine or a placebo in a repeated measures design.

DETAILED DESCRIPTION:
This study seeks to determine whether a simple, single intervention of Cetirizine / Zyrtec® use can improve exercise performance of active individuals when acutely exposed to altitude. For this project, healthy subjects will perform steady state and progressive work rate exercise, endurance performance time trials, and repeated sprint performance time trials in the laboratory at a simulated altitude of 3000m (9900ft) after dosing with 10 mg of Cetirizine or a placebo in a repeated measures design. Non-invasive techniques (pulse oximetry, near-infrared spectroscopy [NIRS]) will be utilized to measure changes in arterial oxyhemoglobin saturation and skeletal muscle oxygenation at the level of the microvasculature during exercise. It is expected that after Cetirizine, blood and muscle microvascular oxygenation during heavy exercise will improve compared to placebo, ultimately improving exercise performance at altitude. Subjects will be asked to report to the laboratory on a three occasions, separated by a minimum of 48 hours and a maximum of 14 days. For each subject, all testing sessions will be performed at the same time of day. Prior to each testing session, subjects will be asked to abstain from caffeine consumption for 12 hours. Subjects will also be asked to avoid alcohol consumption for 24 hours before testing, be at least 3-hour post prandial and avoid high-intensity exercise during the 24 hours leading to the exercise testing. Finally, subjects will be asked to consume a similar diet the night before, and the morning of, Sessions 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Physically active a minimum of 120 minutes a week, as determined by questionnaire
* 18-35 years of age
* Classified as low risk, based on the modified PAR-Q questionnaire, BMI, and non-smoking status
* No history of pulmonary disease and pulmonary function classified as normal, as defined by the following measurements being 80% of predicted values: forced vital capacity (FVC), forced expired volume in one second (FEV1) and FEV1/FVC, according to the American Thoracic Society standards.

Exclusion Criteria:

* Current smoker
* Women who are pregnant or could possibly be pregnant
* BMI > 25 kg/m2
* A 'yes' answer to any of the 14 questions on the PAR-Q pre-participation questionnaire
* History of pulmonary disease or <80% of predicted FCV, FEV1 and/or FEV1/FVC.
* A history of renal or liver disease, due to possible interaction effect with Cetirizine
* Currently taking any prescription or over the counter medications for the treatment of allergies, or taking any of the below listed drugs known to have a moderate or higher interaction effect with Cetirizine:

isocarboxazid tranylcypromine bosutinib clobazam crizotinib daclatasvir eliglustat hyaluronidase lomitapide lurasidone ombitasvir/paritaprevir/ritonavir phenelzine ponatinib ritonavir vemurafenib

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chapman, PhD, Principal Investigator — Indiana University School of Public Health
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
No IPD plan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by direct email to the administrators of the Indiana University ROTC program. It was made clear that participation of cadets was voluntary in nature and was not be a requirement of ROTC duties. Active recruitment took place from 08/2017 to 03/2018.
Pre-assignment Details: Enrolled participants were excluded prior to arm/group assignment if they had abnormal pulmonary function, or voluntarily discontinued with study procedures after completing a graded maximal exercise test and familiarization trial of exercise performance tests on a cycle ergometer. Two subjects withdrew prior to initial group assignments.
Groups:
- Cetirizine/Hypoxia, Placebo/Hypoxia, Placebo/Normoxia: During the first visit, subjects orally ingested 10 mg of Cetirizine 60 min before exercising in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  For the second visit, subjects orally ingested a 10 mg gelatin Placebo 60 min before exercising in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  For the third visit, subjects orally ingested a 10 mg gelatin Placebo 60 min before exercising in a normoxic (room-air) environment (20.9% oxygen).
- Placebo/Hypoxia, Placebo/Normoxia, Cetirizine/Hypoxia: During the first visit, subjects orally ingested a 10 mg Placebo 60 min before exercising in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  For the second visit, subjects orally ingested a 10 mg gelatin Placebo 60 min before exercising in a normoxic (room-air) environment (20.9% oxygen).
  For the third visit, subjects orally ingested 10 mg Cetirizine 60 min before exercising in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
- Placebo/Normoxia, Cetirizine/Hypoxia, Placebo/Hypoxia: During the first visit, subjects orally ingested a 10 mg gelatin Placebo 60 min before exercising in a normoxic (room-air) environment (20.9% oxygen).
  For the second visit, subjects orally ingested 10 mg Cetirizine 60 min before exercising in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  For the third visit, subjects orally ingested a 10 mg Placebo 60 min before exercising in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
- Cetirizine/Hypoxia, Placebo/Normoxia, Placebo/Hypoxia: During the first visit, subjects orally ingested 10 mg Cetirizine 60 min before exercising in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  For the second visit, subjects orally ingested a 10 mg gelatin Placebo 60 min before exercising in a normoxic (room-air) environment (20.9% oxygen).
  For the third visit, subjects orally ingested a 10 mg Placebo 60 min before exercising in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
- Placebo/Normoxia, Placebo/Hypoxia, Cetirizine/Hypoxia: During the first visit, subjects orally ingested a 10 mg gelatin Placebo 60 min before exercising in a normoxic (room-air) environment (20.9% oxygen).
  For the second visit, subjects orally ingested a 10 mg Placebo 60 min before exercising in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  During the third visit, subjects orally ingested 10 mg Cetirizine 60 min before exercising in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
- Placebo/Hypoxia, Cetirizine/Hypoxia, Placebo/Normoxia: During the first visit, subjects orally ingested a 10 mg Placebo 60 min before exercising in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  For the second visit, subjects orally ingested 10 mg Cetirizine 60 min before exercising in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  For the third visit, subjects orally ingested a 10 mg gelatin Placebo 60 min before exercising in a normoxic (room-air) environment (20.9% oxygen).
Period: First Intervention (d1)
Arm/Group | Cetirizine/Hypoxia, Placebo/Hypoxia, Placebo/Normoxia | Placebo/Hypoxia, Placebo/Normoxia, Cetirizine/Hypoxia | Placebo/Normoxia, Cetirizine/Hypoxia, Placebo/Hypoxia | Cetirizine/Hypoxia, Placebo/Normoxia, Placebo/Hypoxia | Placebo/Normoxia, Placebo/Hypoxia, Cetirizine/Hypoxia | Placebo/Hypoxia, Cetirizine/Hypoxia, Placebo/Normoxia
Started | 1 | 5 | 2 | 1 | 1 | 1
Completed | 1 | 5 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: First Washout (>6d)
Arm/Group | Cetirizine/Hypoxia, Placebo/Hypoxia, Placebo/Normoxia | Placebo/Hypoxia, Placebo/Normoxia, Cetirizine/Hypoxia | Placebo/Normoxia, Cetirizine/Hypoxia, Placebo/Hypoxia | Cetirizine/Hypoxia, Placebo/Normoxia, Placebo/Hypoxia | Placebo/Normoxia, Placebo/Hypoxia, Cetirizine/Hypoxia | Placebo/Hypoxia, Cetirizine/Hypoxia, Placebo/Normoxia
Started | 1 | 5 | 2 | 1 | 1 | 1
Completed | 1 | 5 | 1 | 1 | 1 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1
Period: Second Intervention (d1)
Arm/Group | Cetirizine/Hypoxia, Placebo/Hypoxia, Placebo/Normoxia | Placebo/Hypoxia, Placebo/Normoxia, Cetirizine/Hypoxia | Placebo/Normoxia, Cetirizine/Hypoxia, Placebo/Hypoxia | Cetirizine/Hypoxia, Placebo/Normoxia, Placebo/Hypoxia | Placebo/Normoxia, Placebo/Hypoxia, Cetirizine/Hypoxia | Placebo/Hypoxia, Cetirizine/Hypoxia, Placebo/Normoxia
Started | 1 | 5 | 1 | 1 | 1 | 0
Completed | 1 | 5 | 1 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Washout (>6d)
Arm/Group | Cetirizine/Hypoxia, Placebo/Hypoxia, Placebo/Normoxia | Placebo/Hypoxia, Placebo/Normoxia, Cetirizine/Hypoxia | Placebo/Normoxia, Cetirizine/Hypoxia, Placebo/Hypoxia | Cetirizine/Hypoxia, Placebo/Normoxia, Placebo/Hypoxia | Placebo/Normoxia, Placebo/Hypoxia, Cetirizine/Hypoxia | Placebo/Hypoxia, Cetirizine/Hypoxia, Placebo/Normoxia
Started | 1 | 5 | 1 | 1 | 1 | 0
Completed | 1 | 5 | 1 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (d1)
Arm/Group | Cetirizine/Hypoxia, Placebo/Hypoxia, Placebo/Normoxia | Placebo/Hypoxia, Placebo/Normoxia, Cetirizine/Hypoxia | Placebo/Normoxia, Cetirizine/Hypoxia, Placebo/Hypoxia | Cetirizine/Hypoxia, Placebo/Normoxia, Placebo/Hypoxia | Placebo/Normoxia, Placebo/Hypoxia, Cetirizine/Hypoxia | Placebo/Hypoxia, Cetirizine/Hypoxia, Placebo/Normoxia
Started | 1 | 5 | 1 | 1 | 1 | 0
Completed | 1 | 5 | 1 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline characteristics for subjects completing all three study arms (Hypoxia/Cetirizine, Hypoxia/Placebo, Normoxia/Placebo) are included.
Groups:
- Subjects Completing All 3 Study Arms: Completed: Hypoxia/ Cetirizine (14.3% oxygen with 10mg cetirizine), Hypoxia/ Placebo (21% oxygen with gelatin placebo), and Normoxia/Placebo (21% oxygen with gelatin placebo)
Arm/Group | Subjects Completing All 3 Study Arms
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8
Body Fat Percentage [Mean (Standard Deviation); unit: percentage] | 12.1 (3.9)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23 (2)
Maximal Aerobic Capacity (VO2max) [Mean (Standard Deviation); unit: ml/kg/min] | 44.3 (8.3)
Height [Mean (Standard Deviation); unit: cm] | 172 (8)
Weight [Mean (Standard Deviation); unit: kg] | 68.3 (11.1)
Physical Activity [Mean (Standard Deviation); unit: minutes per week] | 441 (310)

OUTCOME MEASURES:

1. Primary Outcome: Performance Time
Description: Time to complete 8km cycling time trial
Time Frame: Performed 60min after pill ingestion
Population: Subjects who completed all three interventions were included in the outcome analysis.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Cetirizine and Hypoxia: 10 mg of Cetirizine given 60 min before exercise in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  Cetirizine: Cetirizine tablet 10 mg
- Placebo and Hypoxia: Placebo given 60 min prior to exercise in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  Placebo oral capsule: Gelatin placebo
- Placebo and Normoxia: Placebo given 60 min prior to exercise in a normobaric room-air environment (21% oxygen).
  Placebo oral capsule: Gelatin placebo
Arm/Group | Cetirizine and Hypoxia | Placebo and Hypoxia | Placebo and Normoxia
Number analyzed (Participants) | 8 | 8 | 8
minutes | 17.03 (1.92) | 18.08 (2.87) | 16.32 (1.98)
Statistical Analysis 1: Comparison: Cetirizine and Hypoxia vs Placebo and Hypoxia vs Placebo and Normoxia; Test type: Superiority; p = 0.047, ANOVA; The overall model was adjusted for the co-variate "VO2max."; Mean Difference (Final Values) = 1.06, 95% CI 2-sided [0.01 to 2.11]

2. Secondary Outcome: Plasma Histamine Concentrations at Baseline and Post-Exercise
Description: Plasma histamine concentrations (ng/mL) were determined baseline and post-exercise for each experimental condition. Baseline measures were taken immediately prior to exercise and the post-exercise measures were taken 5-10 minutes after the cessation of exercise.
Time Frame: baseline and immediately post-exercise, same day as pill ingestion
Population: Subjects included are those who completed all three intervention visits.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cetirizine and Hypoxia (Baseline): 10mg Cetirizine given 60 min prior to exercise in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  Placebo oral capsule: 10 mg Cetirizine Histamine: assessed 60 min after pill ingestion, prior to exercise
- Cetirizine and Hypoxia (Post-Exercise): 10mg Cetirizine given 60 min prior to exercise in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  Placebo oral capsule: 10 mg Cetirizine Histamine: assessed 60 min after pill ingestion, 5-10 min after 8km time trial exercise
- Placebo and Hypoxia (Baseline): Placebo given 60 min prior to exercise in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  Placebo oral capsule: gelatin placebo Histamine: assessed 60 min after pill ingestion, prior to exercise
- Placebo and Hypoxia (Post-Exercise): Placebo given 60 min prior to exercise in a normobaric hypoxic environment (14.3% oxygen simulating an altitude of 3,000m/9,000ft).
  Placebo oral capsule: gelatin placebo Histamine: assessed 60 min after pill ingestion, 5-10 after 8km time trial exercise
- Placebo and Normoxia (Baseline): Placebo given 60 min prior to exercise in a normobaric room-air environment (21% oxygen).
  Placebo oral capsule: gelatin placebo Histamine: assessed 60 min after pill ingestion, prior to exercise
- Placebo and Normoxia (Post-Exercise): Placebo given 60 min prior to exercise in a normobaric room-air environment (21% oxygen).
  Placebo oral capsule: gelatin placebo Histamine: assessed 60 min after pill ingestion, 5-10 min following 8km time trial exercise
Arm/Group | Cetirizine and Hypoxia (Baseline) | Cetirizine and Hypoxia (Post-Exercise) | Placebo and Hypoxia (Baseline) | Placebo and Hypoxia (Post-Exercise) | Placebo and Normoxia (Baseline) | Placebo and Normoxia (Post-Exercise)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
ng/mL | .36 (.14) | .49 (.21) | .56 (.39) | .61 (.34) | .37 (.09) | .47 (.15)
Statistical Analysis 1: Comparison: Cetirizine and Hypoxia (Baseline) vs Cetirizine and Hypoxia (Post-Exercise) vs Placebo and Hypoxia (Baseline) vs Placebo and Hypoxia (Post-Exercise) vs Placebo and Normoxia (Baseline) vs Placebo and Normoxia (Post-Exercise); Test type: Superiority; p = 0.327, ANOVA
Statistical Analysis 2: Comparison: Cetirizine and Hypoxia (Baseline); Test type: Superiority; p = 0.557, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at the time of each intervention visit and for a period of up to one month following each intervention visit date.
Description: The definition of adverse event and/or serious adverse event does not differ from clinicaltrials.gov definitions. All-cause mortality was monitored/assessed.
Arm/Group | Cetirizine and Hypoxia | Placebo and Hypoxia | Placebo and Normoxia
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/11 | 0/11 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetirizine and Hypoxia (N=11) | Placebo and Hypoxia (N=11) | Placebo and Normoxia (N=11)
Fainting (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Lightheadedness and fainting episode with blood draw procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03192488/Prot_SAP_000.pdf